CLINICAL TRIAL: NCT01088828
Title: The Pma Mouse and the Developmental Basis of Clubfoot: MRI Anatomical Modelling of Human ICTEV (Clubfoot)
Brief Title: Exploring the Causes of Clubfoot Using Magnetic Resonance Imaging, MRI
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: MRC/BM056
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Clubfoot
Keywords: MRI, clubfoot, CTEV, Congenital Talipes Equinovarus
MeSH Terms: conditions — Clubfoot | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Group A: Foetuses with clubfoot identified in utero (n=15). Of these:
  * around 10 will be born with clubfoot and will form most of Group B,
  * around 5 will be born without clubfoot and will form part of group C.
  Interventions: Other: Magnetic Resonance Imaging (MRI) of calf and foot
- Group B: Neonates affected by clubfoot (n=10)
  Interventions: Other: Magnetic Resonance Imaging (MRI) of calf and foot
- Group C: Control group of unaffected neonates (n=10)
  Interventions: Other: Magnetic Resonance Imaging (MRI) of calf and foot
- Group D: Young adults having completed treatment (n=5)
  Interventions: Other: Magnetic Resonance Imaging (MRI) of calf and foot
- Group E: Control group of young unaffected adults (n=5)
  Interventions: Other: Magnetic Resonance Imaging (MRI) of calf and foot

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) of calf and foot — Detailed 3-D comparison of MRI scans of children with clubfoot and controls without clubfoot in utero, in untreated infants and in older children who have been treated.
  Other Names: MR scan

SUMMARY:
The purpose of this study is to:

1. compare structural variations observed in the calf and foot of the clubfoot mouse model(pma)with human clubfoot patients antenatally and postnatally;
2. identify features that might be used in future large scale studies to delineate a subtype of human clubfoot associated with lack of response to standard 'Ponseti' manipulation treatments.

DETAILED DESCRIPTION:
Clubfoot is a medical condition of the foot known to doctors as "Congenital Talipes Equinovarus (CTEV)", which affects at least 2 per 1000 Scottish births (ISD data). Affected babies are born with one or both feet in an abnormal position. Treatment with plaster casts, and occasionally with surgery, is necessary to get the foot into a normal position.

We know from our animal and clinical studies and published work that the normal processes of development of the foot continue through pregnancy and postnatally. Clubfoot has never been studied by MRI antenatally in humans, and examination of the foot before birth may offer aetiological clues, not apparent from a single postnatal scan. Additionally, robust information that will help to understand which features of clubfoot in utero predict a truly affected fetus could be very useful for the clinical care of those suspected to be affected at a 20 week scan. This study will provide preliminary data to determine whether the usefulness of MRI in this context should be explored in future studies.

ELIGIBILITY:
Inclusion Criteria:

Group A - pregnancies suspected to be affected by clubfoot on detailed scan. Group B - neonates / infants with clubfoot. Age Preferably under 3 months). Group C - neonates / infants without clubfoot.Preferably under 3 months). Group D- young adults who have undergone treatment for clubfoot and are not undergoing further active treatment. Age range 14-30 years.

Group E - young adults without known lower limb pathology. Age 14-30 years.

Exclusion Criteria:

For all groups the exclusion criteria are any contraindication to MRI scanning.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group A: Pregnant women carrying a foetus with suspected clubfoot. Group B: Neonates affected by clubfoot Group C: Unaffected neonates Group D: Young adults who have undergone treatment for clubfoot Group E: Control group of young unaffected adults
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zosia H Miedzybrodzka, MBChB, PhD, Principal Investigator — University of Aberdeen; Simon L Barker, FRCS, MD, Principal Investigator — NHS Grampian Health Board
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom